CLINICAL TRIAL: NCT00107770
Title: Safety and Dose Escalating Study of Oral Sodium Phenylbutyrate in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Safety Study of Oral Sodium Phenylbutyrate in Subjects With ALS (Amyotrophic Lateral Sclerosis)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Muscular Dystrophy Association (Other)
Responsible Party: Ferrante, Robert - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0015
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Last update posted 2010-01-11 (Estimated); Status verified 2008-10

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; histone deacetylase inhibition; open label; safety study; sodium phenylbutyrate
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — 4-phenylbutyric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): ALS patient
  Interventions: Drug: sodium phenylbutyrate

INTERVENTIONS:
Drug: sodium phenylbutyrate — histone deacteylase inhibitor

SUMMARY:
The purpose of the study is to evaluate the safety of sodium phenylbutyrate (NaPB) treatment in subjects with amyotrophic lateral sclerosis (ALS) and the ability to take this medication without major side effects.

DETAILED DESCRIPTION:
Although it is known that nerve cells die in the brains and spinal cords of patients who have ALS, the cause of the cell death is unknown. There is evidence that this cell death may be caused by changes in DNA, the body's genetic material. Drugs such as sodium phenylbutyrate (NaPB) can increase the expression of genes, block how the motor nerve cells in ALS die, and may prove to be an effective therapy for ALS. NaPB has shown an improvement in survival in mice with conditions similar to ALS.

STUDY DESIGN:

All research participants will take sodium phenylbutyrate for a total of 20 weeks. The dose of medication will be increased every 2 to 4 weeks until a maximum, easily tolerated dose is achieved (study maximum is 21 g/day).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS
* At least 18 years of age
* Women, who can become pregnant, must actively use effective birth control measures

Exclusion Criteria:

* Must not have any other neurological (nervous system) disease

Veterans only are eligible to participate at VA sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2006-11 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 20 weeks

SECONDARY OUTCOMES:
The number of side effects at each dosage, including abnormalities in vital signs, physical examination, blood tests and EKGs, change in vital capacity (breathing function) and ALS functional rating scale
Relationship between blood levels and sodium phenylbutyrate dosage

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ferrante, PhD MSc, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford
Locations (10):
- United States (10):
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - VA Medical Center, Lexington, Lexington, Kentucky
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, Bedford, Massachusetts
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - VA Medical Center, Syracuse, Syracuse, New York
  - VA Medical Center, Durham, Durham, North Carolina
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Pittsburgh Health Care System, Pittsburgh, Pennsylvania
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas